CLINICAL TRIAL: NCT04847622
Title: A Multi-centre, Multi-country Retrospective Cohort Study to Evaluate the Clinical Outcomes in Adults With Covid-19 Who Have Been Treated With Remdesivir.
Brief Title: Study to Evaluate the Clinical Outcomes in Adults With Covid-19 Who Have Been Treated With Remdesivir.
Acronym: 909REM
Status: Completed | Type: Observational
Sponsor: NEAT ID Foundation (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor
Other Study IDs: NEAT ID 909REM
Record Dates: First submitted 2021-03-17; First posted 2021-04-19 (Actual); Results first posted 2024-11-29 (Actual); Last update posted 2024-11-29 (Actual); Status verified 2024-10

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19 | interventions — remdesivir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Target Population: Adults with COVID-19 diagnosed and treated with Remdesivir after Aug 31st2020.
  Interventions: Drug: Remdesivir

INTERVENTIONS:
Drug: Remdesivir — treated with Remdesivir

SUMMARY:
This is a multi-centre, multi-country retrospective cohort study. At least 450COVID-19 cases from up to 20 participating study sites who meet all eligibility criteria will be included in the analysis. Deidentified data will be extracted from electronic medical record (EMR) databases, clinical registries, case series or additional sources from participating sites and countries, and then entered into a structured e-CRF system. addition, each site/country will be surveyed to determine the local standard of care therapy for COVID-19 infection and to determine if standard protocols were/are in place for the use of Remdesivir and if/how the protocols changed over time.

ELIGIBILITY:
Inclusion Criteria:

All Adult participants with COVID-19 confirmed by PCR who meet the following criteria:

* Hospitalised after August 31st,2020
* Receivedat least one dose of Remdesivir(RDV)at anytime during hospitalisation

Exclusion Criteria:

* Received Remdesivir as part of a clinical trial, compassionate use or expanded access program
* Received Remdesivir prior to this admission at any other health facility than the research sites and whose health records are available.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with COVID-19 diagnosed and treated with Remdesivir after Aug 31st2020.
Sampling Method: Non-Probability Sample
Enrollment: 451 (Actual)
Dates: Start 2021-02-12 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (12):
- France (3):
  - CHU de Nantes, Nantes
  - Hospital Lariboisiere, Paris
  - Hopital Saint-Louis, Paris
- Tel Aviv Sourasky Medical Center, Tel Aviv, Israel
- Erasmus Medical Center, Rotterdam, Netherlands
- Spain (5):
  - Hospital Germans Trias i Pujol, Barcelona
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital Universitari Vall d'Herbon, Barcelona
  - Hospital Clinico Universitario San Carlos, Madrid
  - Hospital Universitario 12 de Octubre, Madrid
- United Kingdom (2):
  - Royal Free Hospital, London
  - Chelsea & Westminster Hospital, London

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Arber N, Shah PL, Assoumou L, Rokx C, De Castro N, Bakhai A, Soriano Viladomiu A, Mateu L, Lumbreras C, Estrada V, Curran A, Sellier PO, Duffy A, Fletcher C, Mozaffari E, Haubrich R, Hodgkins P, Pozniak A, Raffi F. Clinical outcomes by supplemental oxygen use in remdesivir-treated, hospitalised adults with COVID-19. Infect Dis Now. 2023 Oct;53(7):104760. doi: 10.1016/j.idnow.2023.104760. Epub 2023 Jul 14. PMID 37454762

RESULTS

PARTICIPANT FLOW:
Groups:
- Cases: Adults with COVID-19 diagnosed and treated with Remdesivir after Aug 31st, 2020.
  1. Hospitalised after August 31st,2020
  2. Received at least one dose of Remdesivir (RDV) at any time during hospitalisation
Period: Overall Study
Arm/Group | Cases
Started | 448
Completed | 448
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Cases
Number analyzed (Participants) | 448
Age, Continuous [Median (Full Range); unit: Years] | 65 [54 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 162
  Male | 286
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White Caucasian | 159
  White Mixed | 24
  Asian | 23
  Black | 12
  Other | 230
Pregnant women, n (%) [Count of Participants; unit: Participants] | 0
Body mass index (BMI, Kg/m²) [Median (Inter-Quartile Range); unit: Kg/m²] | 28.4 [24.9 to 32.2]
Comorbidities [Count of Participants; unit: Participants]
  Comorbidities | 355
  Cardiovascular Disease excluding Hypertension | 115
  Diabetes | 138
  Hypertension | 202
  Asthma | 33
  COPD | 29
  Severe renal disease | 16
  Liver Disease | 9
  HIV Infection | 2
  Chemo/radiotherapy for cancer | 46
  Receiving Immuno-Suppressive Agent (Not for Cancer) | 19
  Obesity | 74
  Dementia | 15
NEWS2 score [Count of Participants; unit: Participants] — NEWS2 is a summary score of six physiological parameters (respiratory rate, oxygen saturation, systolic blood pressure, heart rate, level of consciousness, temperature, and supplemental oxygen dependency) recorded routinely when patients present or are admitted to hospital. These parameters are used to generate a severity score classified as low: aggregate score 0-4, low - medium/medium: score of 3 in any individual parameter/aggregate score 5-6,high: aggregate score 7 or more. A higher score indicates a greater clinical risk. Population: Of the total 448 cases, 391 had sufficient baseline data recorded to enable a NEWS2 score to be calculated and were thus included in this analysis
  Participants
    Low: number analyzed (Participants) | 391
    Low | 145
    Low-medium/Medium: number analyzed (Participants) | 391
    Low-medium/Medium | 146
    High: number analyzed (Participants) | 391
    High | 100
SpO2 (%) [Count of Participants; unit: Participants]
  Low disease severity - No supplemental oxygen | 81
  Medium disease severity - Low flow oxygen | 295
  High disease severity - High flow oxygen | 72
Other Treatment for COVID-19, n (%) [Count of Participants; unit: Participants]
  None | 100
  Corticosteroids | 285
  Tocilizimab /Sarilumab | 18
  Other COVID Treatment Related Drug | 45

OUTCOME MEASURES:

1. Primary Outcome: All Case Mortality by Day 28
Description: Occurrence of death within 28 days.
Time Frame: Day 28
Population: Full population analysis - All enrolled participants who met the eligibility criteria and with data available at baseline will be included in the Full Analysis Population. Disease severity was grouped based on oxygen support requirement at baseline: no supple-mental oxygen (NSO), LFO(≤6 litres (l)/minute), and HFO (>6 l/ minute).
Measure: Number; unit: participants
Groups:
- Overall: Adults with COVID-19 hospitalised between August 31st and December 31st 2020 who received at least one dose of remdesivir.
- Low Disease Severity at Baseline: No supplemental oxygen support (NSO)
- Medium Disease Severity at Baseline: Low to medium disease defined by low flow oxygen support (≤6 litres (l)/minute)
- High Disease Severity at Baseline: High disease severity at baseline defined by high flow oxygen support (>6 litres (l)/minute
Arm/Group | Overall | Low Disease Severity at Baseline | Medium Disease Severity at Baseline | High Disease Severity at Baseline
Number analyzed (Participants) | 448 | 81 | 295 | 72
participants | 52 | 5 | 30 | 17

2. Primary Outcome: Duration of Hopitalisation
Description: Number of hospital discharges by day 28.
Time Frame: Day 28
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Overall | Low Disease Severity at Baseline | Medium Disease Severity at Baseline | High Disease Severity at Baseline
Number analyzed (Participants) | 448 | 81 | 295 | 72
participants | 369 | 69 | 248 | 52

3. Secondary Outcome: Clinical Status Assessed by a 7-point Ordinal Clinical Status Scale
Description: Clinical status assessed by a 7-point ordinal scale on Day 7 7-point ordinary scale:
  1. Death
  2. Hospitalised, on invasive mechanical ventilation or ECMO
  3. Hospitalised, on non-invasive ventilation or high flow oxygen devices
  4. Hospitalised, requiring low flow supplemental oxygen
  5. Hospitalised, not requiring supplemental oxygen -requiring ongoing medical care (COVID-19 related or otherwise)
  6. Hospitalised, not requiring supplemental oxygen -no longer requires ongoing medical care
  7. Not hospitalised A higher score indicates a better outcome
Time Frame: Day 7
Population: Hospitalised adult patients with COVID-19 who received at least one dose of remdesivir during their hospital admission.
Measure: Count of Participants; unit: Participants
Arm/Group | Overall | Low Disease Severity at Baseline | Medium Disease Severity at Baseline | High Disease Severity at Baseline
Number analyzed (Participants) | 448 | 81 | 295 | 72
Participants
  Ordinal Scale 1 | 10 | 2 | 3 | 5
  Ordinal Scale 2 | 13 | 1 | 8 | 4
  Ordinal Scale 3 | 80 | 6 | 45 | 29
  Ordinal Scale 4 | 137 | 28 | 98 | 11
  Ordinal Scale 5 | 70 | 16 | 47 | 7
  Ordinal Scale 6 | 67 | 15 | 44 | 8
  Ordinal Scale 7 | 68 | 13 | 47 | 8

4. Secondary Outcome: Clinical Status Assessed by a 7-point Ordinal Clinical Status Scale on Day 14
Description: 7-point ordinal scale:
  1. Death
  2. Hospitalised, on invasive mechanical ventilation or ECMO
  3. Hospitalised, on non-invasive ventilation or high flow oxygen devices
  4. Hospitalised, requiring low flow supplemental oxygen
  5. Hospitalised, not requiring supplemental oxygen -requiring ongoing medical care (COVID-19 related or otherwise)
  6. Hospitalised, not requiring supplemental oxygen -no longer requires ongoing medical care
  7. Not hospitalised A higher score indicates a better outcome
Time Frame: Day 14
Measure: Count of Participants; unit: Participants
Arm/Group | Overall | Low Disease Severity at Baseline | Medium Disease Severity at Baseline | High Disease Severity at Baseline
Number analyzed (Participants) | 448 | 81 | 295 | 72
Participants
  Ordinal Scale 1 | 36 | 5 | 17 | 14
  Ordinal Scale 2 | 15 | 1 | 13 | 1
  Ordinal Scale 3 | 22 | 5 | 11 | 6
  Ordinal Scale 4 | 44 | 8 | 28 | 8
  Ordinal Scale 5 | 38 | 11 | 26 | 1
  Ordinal Scale 6 | 85 | 11 | 56 | 18
  Ordinal Scale 7 | 206 | 40 | 142 | 24

5. Secondary Outcome: Clinical Severity on Day 7, Day 14 and Day 28 Based on National Early Warning Score 2 (NEWS2) Score
Description: NEWS2 is a summary score of six physiological parameters (respiratory rate, oxygen saturation, systolic blood pressure, heart rate, consciousness, temperature, and supplemental oxygen dependency). The parameters are assessed to generate a severity score classified as low: aggregate score 0-4, low - medium/medium: score of 3 in any individual parameter/aggregate score 5-6,high: aggregate score 7 or more. A higher score indicates a greater clinical risk.
  Clinical status assessed by a 7-point ordinal scale.7-point ordinary scale:
  1. Death
  2. Hospitalised,on invasive mechanical ventilation or ECMO
  3. Hospitalised,on non-invasive ventilation or high flow oxygen devices
  4. Hospitalised,requiring low flow supplemental oxygen
  5. Hospitalised,not requiring supplemental oxygen -requiring ongoing medical care (COVID-19 related or otherwise)
  6. Hospitalised,not requiring supplemental oxygen -no longer requires ongoing medical care
  7. Not hospitalised A higher score indicates a better outcome.
Time Frame: Day 7, 14, and 28
Population: Of the total of 448 hospitalised adult COVID-19 patients who received at least one dose of remdesivir, these 391 (87%) had sufficient baseline data recorded to enable a NEWS2 score to be calculated and were thus included in this analsis
Measure: Count of Participants; unit: Participants
Groups:
- Low Severity: Aggregate Score 0-4
- Low - Medium/ Medium Severity: Score of 3 in any individual parameter
- High Severity: Aggregate score 7 or more
- Overall: All cases
Arm/Group | Low Severity | Low - Medium/ Medium Severity | High Severity | Overall
Number analyzed (Participants) | 145 | 146 | 100 | 391
Participants
  Ordinal Scale 1 at day 7 | 2 | 3 | 4 | 9
  Ordinal Scale 2 at day 7 | 3 | 4 | 4 | 11
  Ordinal Scale 3 at day 7 | 26 | 26 | 24 | 76
  Ordinal Scale 4 at day 7 | 45 | 46 | 28 | 119
  Ordinal Scale 5 at day 7 | 25 | 16 | 14 | 55
  Ordinal Scale 6 at day 7 | 27 | 20 | 12 | 59
  Ordinal Scale 7 at day 7 | 17 | 31 | 14 | 62
  Ordinal Scale 1 at day 14 | 12 | 8 | 13 | 33
  Ordinal Scale 2 at day 14 | 2 | 8 | 3 | 13
  Ordinal Scale 3 at day 14 | 7 | 6 | 6 | 19
  Ordinal Scale 4 at day 14 | 15 | 14 | 10 | 39
  Ordinal Scale 5 at day 14 | 13 | 7 | 5 | 25
  Ordinal Scale 6 at day 14 | 28 | 32 | 21 | 81
  Ordinal Scale 7 at day 14 | 68 | 71 | 42 | 181
  Ordinal Scale 1 at day 28 | 14 | 14 | 19 | 47
  Ordinal Scale 2 at day 28 | 0 | 3 | 1 | 4
  Ordinal Scale 3 at day 28 | 2 | 1 | 2 | 5
  Ordinal Scale 4 at day 28 | 3 | 6 | 3 | 12
  Ordinal Scale 5 at day 28 | 3 | 3 | 1 | 7
  Ordinal Scale 6 at day 28 | 11 | 9 | 7 | 27
  Ordinal Scale 7 at day 28 | 112 | 110 | 67 | 289

6. Secondary Outcome: Clinical Status Assessed by a 7-point Ordinal Clinical Status Scale on Day 28
Description: Clinical status assessed by a 7-point ordinal clinical status scale on Day 28 (or at last observation if discharged or died prior to this time point) in those still hospitalised after Day 14 7-point ordinary scale:
  1. Death
  2. Hospitalised, on invasive mechanical ventilation or ECMO
  3. Hospitalised, on non-invasive ventilation or high flow oxygen devices
  4. Hospitalised, requiring low flow supplemental oxygen
  5. Hospitalised, not requiring supplemental oxygen -requiring ongoing medical care (COVID-19 related or otherwise)
  6. Hospitalised, not requiring supplemental oxygen -no longer requires ongoing medical care
  7. Not hospitalised
Time Frame: Day 28
Population: Hospitalised Adults with COVID-19 who received at least one dose of remdesivir.
Measure: Count of Participants; unit: Participants
Arm/Group | Overall | Low Disease Severity at Baseline | Medium Disease Severity at Baseline | High Disease Severity at Baseline
Number analyzed (Participants) | 448 | 81 | 295 | 72
Participants
  Ordinal Scale 1 | 52 | 5 | 30 | 17
  Ordinal Scale 2 | 4 | 0 | 4 | 0
  Ordinal Scale 3 | 6 | 4 | 0 | 2
  Ordinal Scale 4 | 14 | 1 | 9 | 4
  Ordinal Scale 5 | 8 | 1 | 7 | 0
  Ordinal Scale 6 | 27 | 5 | 15 | 7
  Ordinal Scale 7 | 333 | 64 | 227 | 42

7. Secondary Outcome: SpO2 > 94% on Room Air
Description: Number of participants SpO2 > 94% on room air by day 28
Time Frame: Day 28
Population: Adults with hospitalised COVID-19 who received at least one dose of remdesivir
Measure: Count of Participants; unit: Participants
Arm/Group | Overall | Low Disease Severity at Baseline | Medium Disease Severity at Baseline | High Disease Severity at Baseline
Number analyzed (Participants) | 448 | 81 | 295 | 72
Participants | 154 | 22 | 113 | 19

8. Secondary Outcome: Duration of Oxygen Therapy
Description: Median (IQR) duration on oxygen therapy by day 28.
Time Frame: Day 28
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Overall | Low Disease Severity at Baseline | Medium Disease Severity at Baseline | High Disease Severity at Baseline
Number analyzed (Participants) | 448 | 81 | 295 | 72
days | 6 [4 to 9] | 5 [3 to 8] | 6 [4 to 9] | 6 [4 to 12]

9. Secondary Outcome: ICU Admission
Description: Intensive care unit admission over entire study period
Time Frame: Day 28
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Overall | Low Disease Severity at Baseline | Medium Disease Severity at Baseline | High Disease Severity at Baseline
Number analyzed (Participants) | 448 | 81 | 295 | 72
participants | 55 | 3 | 33 | 19

10. Secondary Outcome: Duration of ICU
Description: Number of days spent in ICU
Time Frame: through study completion, 28 days
Population: Hospitalised Adults with COVID-19 who received at least one dose of remdesivir.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Overall | Low Disease Severity at Baseline | Medium Disease Severity at Baseline | High Disease Severity at Baseline
Number analyzed (Participants) | 448 | 81 | 295 | 72
days | 13 [8 to 19] | 10 [7 to 11] | 17 [10 to 17] | 10 [6 to 16]

11. Secondary Outcome: Mechanical Ventilation/ECMO Use
Description: Use of mechanical ventilation/ECMO (extracorporeal membrane oxygenation) over study period
Time Frame: Day 28
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Overall | Low Disease Severity at Baseline | Medium Disease Severity at Baseline | High Disease Severity at Baseline
Number analyzed (Participants) | 448 | 81 | 295 | 72
participants | 25 | 3 | 17 | 5

12. Secondary Outcome: Timing of Remdesivir Exposure
Description: Median (IQR) time from first symptoms to use of remdesivir
Time Frame: Day 28
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Overall | Low Disease Severity at Baseline | Medium Disease Severity at Baseline | High Disease Severity at Baseline
Number analyzed (Participants) | 448 | 81 | 295 | 72
days | 7 [4 to 9] | 7 [4 to 11] | 7 [4 to 9] | 7 [5 to 9]

13. Secondary Outcome: Timing From Hospitalisation to Remdesivir Exposure
Description: Median (IQR) time from hospitalisation to use of remdesivir
Time Frame: Day 28
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Overall | Low Disease Severity at Baseline | Medium Disease Severity at Baseline | High Disease Severity at Baseline
Number analyzed (Participants) | 448 | 81 | 295 | 72
days | 1 [0 to 2] | 2 [1 to 3] | 1 [0 to 2] | 1 [0 to 1]

14. Secondary Outcome: Duration of Remdesivir Use
Description: Median (IQR) duration of use of remdesivir
Time Frame: Day 28
Population: as for outcome 1
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | Overall | Low Disease Severity at Baseline | Medium Disease Severity at Baseline | High Disease Severity at Baseline
Number analyzed (Participants) | 448 | 81 | 295 | 72
days | 5 [4 to 5] | 5 [4 to 6] | 5 [4 to 5] | 5 [3 to 6]

15. Secondary Outcome: Readmission With COVID-19 Complications
Description: Re-admission with COVID-19 complications or recurrence within 28 days of discharge and outcome
Time Frame: Day 28
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Overall | Low Disease Severity at Baseline | Medium Disease Severity at Baseline | High Disease Severity at Baseline
Number analyzed (Participants) | 448 | 81 | 295 | 72
Participants | 16 | 3 | 11 | 2

ADVERSE EVENTS:
Time Frame: Day 28
Description: All cause mortality was collected throughout the study period. All other adverse events (not including all cause mortality) were not collected.
Groups:
- Control Group: Adults with COVID-19 diagnosed and treated with Remdesivir after Aug 31st 2020.
Arm/Group | Control Group
All-Cause Mortality (participants affected / at risk) | 52/448
Serious Adverse Events (participants affected / at risk) | 52/448
Other Adverse Events (participants affected / at risk) | 0/0
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control Group (N=448)
Mortality (Respiratory, thoracic and mediastinal disorders) | 52 (52)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-12-17): https://cdn.clinicaltrials.gov/large-docs/22/NCT04847622/Prot_000.pdf
  • Statistical Analysis Plan (2021-05-07): https://cdn.clinicaltrials.gov/large-docs/22/NCT04847622/SAP_001.pdf